CLINICAL TRIAL: NCT05402956
Title: Effect of Aerobic Exercise Training in Persons With Multiple Sclerosis With Restless Legs Syndrome
Brief Title: Aerobic Exercise in Persons With Multiple Sclerosis With Restless Legs Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, PhD, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/12-18
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental)
  Interventions: Behavioral: Aerobic exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Aerobic exercise — Moderate aerobic exercise training
  Arms: Aerobic exercise

SUMMARY:
In this studly, the effects of an 12-week aerobic exercise training in persons with multiple sclerosis with restless legs syndrome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* A relapsing-remitting or secondary progressive type of multiple sclerosis,
* To be willing to participate in the study.

Exclusion Criteria:

* Another neurological disorder,
* Orthopedic surgery history including the ankle-foot, knee, hip, or spine, affecting balance,
* Diagnosed severe cognitive and/or psychiatric impairment,
* Having congestive heart failure, coronary, cerebrovascular, and pulmonary disease such as COPD
* Having cardiac disease such as hypertension that would be a contraindication to exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group rating scale for restless legs syndrome | Change from Baseline at 12 weeks
  The International Restless Legs Syndrome Study Group rating scale for restless legs syndrome is used to assess severity of the restless legs syndrome symptoms. It consists of 10 items scored by 0 to 4. Possible scores range from 0 to 40. Higher scores indicate higher severity.

SECONDARY OUTCOMES:
Timed 25-Foot Walk | Change from Baseline at 12 weeks
  The Timed 25-Foot Walk is a quantitative mobility and leg function performance test based on a timed 25-walk. he patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score is the average of the two completed trials. Higher time represents slower walking speed and more walking impairment.
12-Item Multiple sclerosis walking scale | Change from Baseline at 12 weeks
  The 12-Item Multiple sclerosis walking scale is a self-assessment scale which measures the impact of multiple sclerosis on walking. It consists of 12 questions with Likert-type choose options concerning the limitations to walking due to multiple sclerosis during the past 2 weeks. Total score ranges 0 from 100. Higher scores indicate more impact of multiple sclerosis on walking.
Epworth Sleepiness Scale | Change from Baseline at 12 weeks
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Multiple Sclerosis International Quality of Life questionnaire | Change from Baseline at 12 weeks
  The Multiple Sclerosis International Quality of Life questionnaire is a disease-specific, self-administered, multidimensional questionnaire, was co-developed and initially validated in 15 countries including Turkey. The questionnaire comprises 31 questions in 9 subscales: activities of daily living, psychological well-being, symptoms, relationships with friends, relationships with family, sentimental and sexual life, coping, rejection, and relationships with healthcare system. All 9 dimensions and the index score were linearly transformed and standardized on a 0-100 scale, where 0 indicates the worst possible level of quality of life and 100 indicates the best level.
Pittsburgh Sleep Quality Index | Change from Baseline at 12 weeks
  Detect sleep disturbances or deficits.
Time Up and Go Test | Change from Baseline at 12 weeks
  Assessments will be performed with APDM Opals.
Six-Minute Walk Test | Change from Baseline at 12 weeks
  The 6-Minute Walk Test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The goal is for the individual to walk as far and fast as possible in 6 minutes. The total distance is recorded. Higher distance represents a better submaximal exercise capacity.
Two-Minute Walk Test | Change from Baseline at 12 weeks
  Assessments will be performed with APDM Opals.
Estimated VO2 Max | Change from Baseline at 12 weeks
  Estimated VO2max will be calculated Astrand-Rhyming Cycle Ergometer Test.

OTHER OUTCOMES:
Restless Legs Syndrome Diagnostic Criteria | At Baseline
  Diagnostic Criteria for Restless Legs Syndrome was developed by the Restless Legs Syndrome Working Group in 1995 and revised in 2003 and 2014. These criteria include; the need to move the legs due to uncomfortable or unpleasant sensations in the legs, the need for movement or disturbing sensations start or worsen at rest, the need for movement or disturbing sensations can be partially or totally relieved by movements such as walking or stretching, the need for movement or disturbing sensations may worsen at night or only occur in the evening or night, The aforementioned features cannot be considered only in relation to primary symptoms or other medical or behavioral conditions (e.g., myalgia, venous stasis, leg edema, leg cramps, habitual foot swing). Patients meeting all of the criteria are diagnosed with restless legs syndrome. The restless legs syndrome diagnosis will be confirmed by a neurologist.
Expanded Disability Status Scale | At Baseline
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale is based on a neurological examination by a clinician. It has steps from 0 to 10. The higher scores indicate higher neurological disability

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Hospital, MS Outpatient Clinic, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided